CLINICAL TRIAL: NCT05203198
Title: Primary Care Based Depression Prevention in Adolescents: Intervention Optimization in Preparation for Implementation Study
Brief Title: The PATHway Study: Primary Care Based Depression Prevention in Adolescents
Acronym: PATHway
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Wake Forest University Health Sciences (Other); Endeavor Health (Other); University of Chicago (Other); National Institute of Mental Health (NIMH) (NIH); Mile Square Health Center (Other); Lawndale Christian Health Center (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Benjamin Van Voorhees, MD, MPH, Professor and Head, Department of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: CHAIRb 20080601; 1R01MH124723-01 (NIH); 3R01MH124723-04S1 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Depression; Mental Disorder in Adolescence
Keywords: Adolescents Depression; Internet intervention; Cognitive-Behavioral Therapy; Prevention; MOST design
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: The Multiphase Optimization Strategy (MOST) will be utilized to optimize a primary care, technology-based intervention (CATCH-IT) for the prevention of depression in at-risk adolescents to optimize efficacy, tolerability and scalability for implementation studies and eventual dissemination. This MOST process includes: (1) theoretical organization of components, target behaviors and links to preventive outcomes (vulnerability and protective factors, likelihood of developing depressive episode), (2) selection of components for factorial design, (3) optimization criteria and (4) factorial design (randomization, intervention delivery, assessments, analysis and optimization). The theoretically grounded components selected are: (1) behavioral activation modules; (2) cognitive-behavioral therapy modules; (3) interpersonal psychotherapy modules; and (4) parent program modules.
Who Masked: Outcomes Assessor
Masking Description: Subjects will know the condition to which they are randomized when opening their CATCH-IT login, as the number of components will be apparent on the sidebar of the webpage.
  All clinical evaluators conducting the MINI Kid and other psychological assessments will work out of the Boston Call Center and they will be the only staff blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- 1. No adolescent modules + no parent modules (No Intervention): No adolescent nor parent modules will be offered to the participant.
- 2. Adolescent behavioral activation modules only (Experimental): Adolescent behavioral activation modules only
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 3. Adolescent cognitive-behavioral therapy modules only (Experimental): Adolescent cognitive-behavioral therapy modules only
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 4. Adolescent interpersonal therapy modules only (Experimental): Adolescent interpersonal therapy modules only
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 5. Adolescent behavioral activation modules + cognitive-behavioral therapy modules (Experimental): Adolescent behavioral activation modules Adolescent cognitive-behavioral therapy modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 6. Adolescent behavioral activation modules + interpersonal therapy modules (Experimental): Adolescent behavioral activation modules Adolescent interpersonal therapy modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 7. Adolescent cognitive-behavioral therapy modules + interpersonal therapy modules (Experimental): Adolescent cognitive-behavioral therapy modules Adolescent interpersonal therapy modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 8. Full Adolescent program only (Experimental): Adolescent behavioral activation modules Adolescent cognitive-behavioral therapy modules Adolescent interpersonal therapy modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 9. Parent program modules only (Experimental): Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 10. Adolescent behavioral activation modules + parent program modules (Experimental): Adolescent behavioral activation modules Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 11. Adolescent cognitive-behavioral therapy modules + parent program modules (Experimental): Adolescent cognitive-behavioral therapy modules Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 12. Adolescent interpersonal therapy modules + parent program modules (Experimental): Adolescent interpersonal therapy modules Parent Program
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 13. Adolescent behavioral activation + cognitive-behavioral therapy + parent program modules (Experimental): Adolescent behavioral activation modules Adolescent cognitive-behavioral therapy modules Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 14. Adolescent behavioral activation + interpersonal therapy + parent program modules (Experimental): Adolescent behavioral activation modules Adolescent interpersonal therapy modules Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 15. Adolescent cognitive-behavioral therapy + interpersonal therapy + parent program modules (Experimental): Adolescent cognitive-behavioral therapy modules Adolescent interpersonal therapy modules Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training
- 16. All adolescent + parent program modules (Active Comparator): Adolescent behavioral activation modules Adolescent cognitive-behavioral therapy modules Adolescent interpersonal therapy modules Parent program modules
  Interventions: Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training

INTERVENTIONS:
Behavioral: Competent Adulthood Transition with Cognitive-Behavioral, Humanistic and Interpersonal Training — Self-directed, technology-based, depression prevention program for adolescents and parents.
  Other Names: CATCH-IT
  Arms: 10. Adolescent behavioral activation modules + parent program modules; 11. Adolescent cognitive-behavioral therapy modules + parent program modules; 12. Adolescent interpersonal therapy modules + parent program modules; 13. Adolescent behavioral activation + cognitive-behavioral therapy + parent program modules; 14. Adolescent behavioral activation + interpersonal therapy + parent program modules; 15. Adolescent cognitive-behavioral therapy + interpersonal therapy + parent program modules; 16. All adolescent + parent program modules; 2. Adolescent behavioral activation modules only; 3. Adolescent cognitive-behavioral therapy modules only; 4. Adolescent interpersonal therapy modules only; 5. Adolescent behavioral activation modules + cognitive-behavioral therapy modules; 6. Adolescent behavioral activation modules + interpersonal therapy modules; 7. Adolescent cognitive-behavioral therapy modules + interpersonal therapy modules; 8. Full Adolescent program only; 9. Parent program modules only

SUMMARY:
Prevention of depressive disorders has become a key priority for the NIMH, but the investigators have no widely available public health strategy to reduce morbidity and mortality. To address this need, the investigators developed and evaluated the primary care based-technology "behavioral vaccine," Competent Adulthood Transition with Cognitive-Behavioral Humanistic and Interpersonal Therapy (CATCH-IT). The investigators will engage N=4 health systems representative of the United States health care system, and conduct a factorial design study to optimize the intervention in preparation for an implementation study and eventual dissemination.

DETAILED DESCRIPTION:
With more than 13% of adolescents diagnosed with depressive disorders each year, prevention of depressive disorders has become a key priority for the National Institute of Mental Health (NIMH). Unfortunately, the investigators have no widely available interventions to reduce morbidity and mortality (e.g. public health impact). To address this need, the investigators developed a multi-health system "collaboratory" to develop and evaluate the primary care based technology "behavioral vaccine," Competent Adulthood Transition with Cognitive-Behavioral Humanistic and Interpersonal Therapy (CATCH-IT) (14 adolescent, 5 parent modules). Using this health-system collaboratory model, the full CATCH-IT program (all modules), demonstrated evidence of efficacy in prevention of depressive episodes in phase-three clinical trials in the United States and China. However, like many "package" interventions, CATCH-IT became larger and more complex across efficacy trials. Thus, adolescents were less willing to complete all 14 modules, suggesting adolescent dose "tolerability" issues (e.g., satisfaction, acceptability and resource use, "time as cost"). Similarly, primary care practices have "scalability" challenges (acceptability, feasibility, resource use, cost), resulting in declining REACH (percent of at-risk youth who complete intervention). To prepare for implementation studies and dissemination, the investigators need to address adolescent tolerability and practice/health system scalability, while preserving efficacy. Multiphase Optimization Strategy (MOST) uses a systematic analytic approach and a factorial randomized clinical trial design to address efficacy, tolerability, and scalability, simultaneously. The investigators will use a MOST approach to optimize CATCH-IT for the prevention of depression (indicated prevention, i.e., elevated symptoms of depression) in practices and health systems representative of US geography and population. The theoretically grounded components of CATCH-IT selected for study and optimization include: behavioral activation, cognitive-behavioral therapy, interpersonal psychotherapy, and parent program. The investigators will use a 4-factor (2x2x2x2) fully crossed factorial design with N=16 cells (25 per cell, 15% dropout) to evaluate the contribution of each component. The investigators propose to randomize N=400 adolescents from multiple sites: Advocate-Aurora Health Care (n=200); Lurie Children's Hospital (n=70); NorthShore University HealthSystem (n=70); University of Chicago Comer Hospital (n=25); University of Texas (n=20); University of Illinois College of Medicine Peoria (n=15). The at-risk youth will be high school students 13 through 18 years old, not currently experiencing a mood disorder, but with subsyndromal symptoms of depression (moderate to high risk). Using the efficient factorial design, the investigators can assess the contribution to prevention efficacy of each component. Thus, the MOST study design will enable us to eliminate non-contributing components while preserving efficacy and to optimize CATCH-IT by strengthening tolerability and scalability by reducing "resource use." By reducing resource use, the investigators anticipate satisfaction and acceptability will also increase, preparing the way for an implementation trial and eventual US Preventive Services Task Force endorsement to support dissemination. Thus, the primary question is whether one component, or perhaps two, can demonstrate an equivalent effect to combinations of other components in terms of efficacy, whilst also demonstrating superior adolescent/family tolerability scalability over a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 13 through 18 years, and
* Adolescents must be experiencing an elevated level of depressive symptoms (PHQ-9 = 5-18), and
* Adolescents will be included if they have had past depressive episode/s, but not if they are in a current depressive episode.

Exclusion Criteria:

1. Outside age range:

   1. 12 or younger
   2. 19 or older
2. Adolescent is a non-English speaker/reader
3. On the PHQ-9 screening, depression symptom level is:

   1. PHQ-9 = 4 or lower
   2. PHQ-9 =19 or higher
4. As assessed by the MINI Kid, a current depressive episode
5. As assessed by the MINI Kid, adolescent meets DSM-5 criteria for a psychotic or bipolar disorder.
6. Currently using medication therapy for depression, anxiety, or other internalizing disorders.
7. Currently engaged in individual treatment for a mood disorder (assessed by BCC during phone screen)
8. Currently engaged in a cognitive-behavioral group or therapy (assessed by BCC during phone screen)
9. Any past psychiatric hospitalizations
10. Any past suicide attempt or incident of self-harm with moderate or greater lethality
11. Extreme, current drug/alcohol abuse (determined by clinician follow up following a score of 3 or greater on the CRAFFT)
12. Current suicidal thoughts

    1. Eligibility will be determined on a case-by-case basis during the baseline PhQ-9 and MINI Kid assessment process and after a consultation with a licensed mental health clinician has taken place. If adolescent report suicidal ideation on the baseline PhQ-9, and found ineligible, the MINI Kid assessment may not be required.
    2. Adolescents with current (within the past 6 months), active suicidal feelings will be excluded.
    3. Adolescents with passive thoughts of death or suicide but report to the mental health clinician that they would never act on these thoughts may be admitted, depending on the severity of the risk.
    4. Adolescents with past (greater than 6 months ago) ideation who are determined to be low risk will be admitted into the study if there has never been an attempt of moderate or greater lethality.
13. Significant reading impairment (a minimum sixth-grade reading level based on parental report) and/or significant intellectual or developmental disabilities
14. Not willing to comply with the study protocol
15. Did not complete phone assessment with MINI Kid by BCC
16. Not affiliated with any of the sites listed in Appendix A.
17. Parent/guardian does not speak English or Spanish
18. Parent/guardian has a cognitive or intellectual impairment
19. Participant Declined/Changed Mind/Uninterested in participating

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Time | Baseline through 12 months
  Time will be measured to nearest minute for all intervention related activities including initial screening, engagement phone calls, use of CATCH-IT. Time will be measured from adolescent, family, practice, community center, healthcare organization, health system perspective. For time that cannot be directly measured by study staff, the investigators will sample direct observation or questionnaires to capture time required for health system related activities such as screening and engagement.
Cultural acceptability adolescent and family | Baseline through 12 months
  Cultural acceptability for each stakeholder using appropriate, validated instruments. Adolescent and family: Usefulness, Satisfaction, and Ease Questionnaire (USE, 30 items, self-report, 7-point Likert scale, 30-210 score range, higher score indicates more acceptable). An example statement is: "I would recommend this to a friend."
Cost | Baseline through 12 months
  Costs will be measured for all stakeholders. For practice, community center, healthcare organizations, health systems, cost will be measured to nearest dollar by converting time measures into employment related costs based on mean wages and benefits for staff at that occupational level. Adolescent and family costs will be measured by converting time into mean hourly wages and benefits for adolescent and family members involved in the project (based on mean wage for age and occupation).
Depressive Symptoms | Baseline through 12 months
  Patient Health Questionnaire-Adolescent (PHQ-A, 9 items plus 4 follow-up items, self-report, 3-point Likert scale, 0-27 score range, higher score indicates more depression symptoms/severity).
Depressive and mental disorder episodes | Baseline through 12 months
  Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI Kid, self-report). This is a structured psychiatric interview administered by a trained staff member which uses stem questions and follow-ups to determine the presence of symptoms and date of onset. The staff member then determines if and when the symptoms developed an episode is present. Measure is either episode present or not and date of onset.
Stress symptoms | Baseline through 12 months
  Center for Epidemiological Studies-Depression Scale (CES-D, 20 items, self-report, measured in frequency, 0,"not at all" to 3, "nearly every day in last week, 0-60 score range, higher score indicates more depressed).
Resiliency | Baseline through 12 months
  Resiliency will be measured across multiple domains. To assess resiliency in terms of coping skills, the Connor-Davidson Resilience Scale (CD-RISC, 10 items, self-report, 4 levels of response, 0-40 score range, higher score indicates better coping skills).
Function | Baseline through 12 months
  Social Adjustment Scale Self-Report (SAS-SR, 23-items, self-report, 5-point Likert scale, 23-115 score range, higher score indicates higher levels of social adjustment) administered to adolescents only.
Relationships (Life Events) | Baseline through 12 months
  University of California at Los Angeles (UCLA) Life Events Scale (19-items, self-report) administered to adolescents only.
Socio-cultural Relevance | Baseline through 12 months
  The Socio-Cultural Relevance Scale (10-item and 14-item versions, self-report, 5-point Likert scale, 10-40 or 14-56 score ranges, higher score indicates greater socio-cultural relevance) will assess perceived change and satisfaction with the intervention, component of cultural acceptability to adolescent)
Acceptability of Intervention | Start to end of recruitment, 32 months
  Acceptability of Intervention Measure (AIM, 1 question with 4 items, self-report, 5-point Likert scale, 1-5 score range, higher score indicates greater acceptability of intervention, to be completed by all staff and leadership, repeatedly, component of cultural acceptability to practice, community center, healthcare organizations, health systems).
Feasibility of Intervention | Start to end of recruitment, 32 months
  Feasibility of Intervention Measure (FIM, 1 question with 4 items, self-report, 5-point Likert scale, 1-5 score range, higher score indicates greater feasibility of intervention, to be completed by all staff and leadership, repeatedly, component of cultural acceptability to practice, community center, healthcare organizations, health systems).
Intervention Appropriateness | Start to end of recruitment, 32 months
  Intervention Appropriateness Measure (IAM, 1 question with 4 items, self-report, 5-point Likert scale, 1-5 score range, higher score indicates greater appropriateness of intervention, to be completed by all staff and leadership, repeatedly, component of cultural acceptability to practice, community center, healthcare organizations, health systems).
Externalizing Behavior Symptoms | Baseline through 12 months
  Disruptive Behavior Disorders Rating Scale-Adolescent (DBD-A, 41-items, self-report, 4-point Likert scale, 0-123 score range, higher score indicates greater externalizing symptoms).
Anxiety Symptoms | Baseline through 12 months
  Screen for Child Anxiety Related Disorders (SCARED, 41-items, self-report, 3-point Likert scale, 0-82 score range, higher score indicates greater anxiety symptoms).
Substance Abuse Symptoms | Baseline through 12 months
  Car, Relax, Alone, Forget, Friends, Trouble substance use assessment (CRAFFT, 6 items, self-report, 2-point scale, 0-6 score range, higher score indicates greater substance abuse symptoms).
Post Traumatic Stress Disorder Symptoms | Baseline through 12 months
  Child Post Traumatic Symptoms Disorder Scale (24-items, self-report, 4-point Likert scale, 0-72 score range, higher score indicates greater PTSD symptom levels).
Rumination | Baseline through 12 months
  Tendency towards rumination will be assessed by the Children's Response Style Scale (CRSS, 10-items, self-report, 5-point Likert scale, 0-50 score range, higher score indicates greater rumination (more repeated negative thinking, less resilient, component of resiliency).
Dysfunctional Attitudes | Baseline through 12 months
  The Dysfunctional Attitude Scale (DAS, 9-item, self-report, 7-point Likert scale, 9-63 score range, higher score indicates more dysfunctional attitude, less resiliency, component of resiliency).
Family Relationships | Baseline through 12 months
  Child Report of Parental Behavior Inventory (CRPBI, 30-item, self-report, 3-point Likert scale, 0-60 score range, higher scores indicate more positive parent child relationship).
Cognitive Style | Baseline through 12 months
  The Children's Cognitive Style Questionnaire (CCSQ, 6-items, self-report, 5-point Likert scale, 0-150 range, higher score indicates greater negativity of cognitive style).
Self-efficacy | Baseline through 12 months
  The Trans-Theoretical Model Scale (TTMS, 10-item, self-report, 4-point Likert scale, 0-24 range, higher score indicates higher self-efficacy and intention to reduce depressive symptoms).
Social Adjustment | Baseline through 12 months
  The Social Adjustment Scale-Adolescent version (SAS-SR, 23-item, self-report, 5-point Likert scale, 0-115 range, higher score indicates higher level of social dysfunction).
Systolic and diastolic blood pressure | At baseline
  Measured in millimeters of mercury.
Height | At baseline
  Measure by standard medical office practice measure, without shoes, in centimeters.
Weight | At baseline
  Measured in kilograms by standard medical office scale, fully clothed participant.
Body Mass Index | At baseline
  Calculated by measuring height (centimeters) and weight (kilogram) to calculate kg/meters squared (BMI, Body Mass Index).

SECONDARY OUTCOMES:
Moderation of COVID-19-related behaviors and consequences | Baseline through 12 months
  The investigators will examine COVID-19-related behaviors and consequences (e.g. social distancing, sheltering-in-place, family illness and death) that that may be moderators of study outcomes using the Holliston at-Home Questionnaire (a 40-item, adolescent self-report, 5-point Likert scale, 0-150 score range, higher score indicates greater behaviors and consequences).
Moderation of COVID-19-related social determinants of health | Baseline through 12 months
  The investigators will examine COVID-19-related social determinants of health (e.g. food insecurity, internet access, unemployment) that may be moderators of study outcomes using the Holliston at-Home Questionnaire (a 40-item, adolescent self-report, 5-point Likert scale, 0-150 score range, higher score indicates greater number of social determinants).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Voorhees, MD, MPH, Principal Investigator — UIC, College of Medicine; Tracy RG Gladstone, PhD, Principal Investigator — Wellesley College; Calvin Rusiewski, MBBS, Study Director — UIC, College of Medicine
Locations (6):
- United States (6):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - UI Health, Chicago, Illinois
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Northshore University HealthSystem, Glenview, Illinois
  - Advocate Aurora Health, Park Ridge, Illinois
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.pathwaystudy.info/